CLINICAL TRIAL: NCT00731575
Title: Viral Inception of Asthma: Prospective Study From Infancy to School-age.
Acronym: VINKU2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Turku (Other)
Collaborators: Cultural Foundation of Finland, Helsinki, Finland (Unknown); Maud Kuistila Foundation, Helsinki, Finland (Unknown); Foundation for Paediatric Research, Finland (Other); Foundation for outpatient Research, Helsinki, Finland (Unknown); Turku University Hospital (Other Government); The Paulo Foundation (Other); Juselius Foundation, Helsinki, Finland (Unknown)
Responsible Party: Tuomas Jartti, Dept of Pediatrics, Turku University Hospital, Turku, Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VINKU2
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Asthma
Keywords: asthma; child; pathogenesis; rhinovirus; prednisolone; Prevention; pediatric
MeSH Terms: conditions — Asthma | interventions — Prednisolone; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: prednisolone — First dose 2 mg/kg (max 60 mg) p.o., then 2 mg/kg/d (max 60 mg/d) p.o. in 3 divided doses for 3 days.
  Other Names: Prednisolon®, 5 mg tablets, Oy Leiras Finland Ab, Helsinki, Finland.

SUMMARY:
The purpose of this study is to study prospectively the early clinical and immunological events in children susceptible to rhinovirus induced early wheezing (i.e., recently found highest risk factor for recurrent wheezing/asthma) and the efficacy of systemic corticosteroid to modify these events.

Up to 50% of children suffer from acute wheezing before school-age. The prevalence of childhood asthma is 5-7%. Although pediatric asthma is mainly allergic, the exacerbations are associated with respiratory viral infections in 95% of cases. The means to predict asthma from environmental factors have been limited mainly to sensitization to aeroallergens (3-fold risk), which start to develop usually at 2-3 years of age. VINKU 1-study (orig. VINKU-study) discovered simultaneously with two other groups, that early wheezing associated with rhinovirus, the "common cold" virus, is the strongest predictor of recurrent wheezing/asthma (up to 10-fold risky). Noteworthily, viral infections work as risk markers already during infancy, a lot earlier than the sensitization to aeroallergens. The investigators also found retrospectively that early wheezers affected by rhinovirus responded to 3 day course of oral prednisolone (inexpensive and widely available treatment): recurrent wheezing decreased by 50% during following 12 months and the difference appeared to continue. VINKU 5V-study is currently investigating the clinical history, prevalence of asthma and airway hyperreactivity of these same children at school-age. The mechanism of rhinovirus associated risk or why they respond to prednisolone are largely unknown. However, the susceptibility to rhinovirus infections is associated with atopy and therefore it is possible these children may have impaired anti-inflammatory (Treg) responses and more likely to wheeze with any pro-inflammatory response (Th1 or Th2). Moreover, they may not effectively clear viruses, because they can not limit rhinovirus to nose and it spreads to lower airways and causes wheezing. VINKU 2-study will prospectively investigate the immunological events in young first-time wheezers affected by rhinovirus, and prospectively study the clinical efficacy of systemic corticosteroid in them. Most likely these children will benefit from the drug in terms of less recurrent wheezing, the investigators will also explore immunological effects of the drug and their link to clinical efficacy. The results are expected to give basis for the prevention of asthma and for the development of new treatment strategies and they can be directly applied to clinical medicine.

DETAILED DESCRIPTION:
Main Hypothesis and Anticipated Results

Virology

1. Rhinovirus is a common causative agent of bronchiolitis.
2. Persistence of rhinovirus (or any virus) infection worsens long-term outcome.
3. The dose of virus inoculation at the time of acute wheezing (assessed semi-quantitatively for rhinovirus and respiratory syncytial virus) is related to outcome.

   Immunology
4. Children susceptible to rhinovirus induced early wheezing have altered immunology (T cell regulation and interferon responses) when compared to children with RSV induced wheezing and children with rhinovirus induced upper respiratory infection without wheezing.
5. These immunological events are related to recurrent wheezing and asthma inception.

   Therapeutic intervention with systemic corticosteroid

   Systemic corticosteroid in children susceptible for rhinovirus-induced early wheezing
6. decreases persistence of rhinovirus infection
7. decreases the severity and relapses of the first wheezing episode, and prevents recurrent wheezing, and asthma,
8. prevents Th2-polarization, favours Th1- and Treg-responses during the treatment period.

Design and Time

Prospective, randomized, double blind, placebo controlled, parallel, one-center trial. The study was commenced in 6/2007.

Inclusion Criteria

Age 3-23 months, be delivered at >37 weeks, first wheezing episode, written informed consent from guardian.

Inclusion Criteria for the Intervention and the Follow-up

Rhinovirus PCR positive wheezing episode and still signs of lower respiratory symptoms (cough, noisy breathing or wheezing) at the time the initiation of study drug.

Inclusion Criteria for the Follow-up without Intervention

Any rhinovirus negative wheezing episode.

Exclusion Criteria

Chronic illness other than atopy, previous systemic or inhaled corticosteroid treatment, participation to another study (excluding long-term follow-up studies in childhood), varicella contact if previously intact, need for intensive care unit treatment, or poor understanding of Finnish.

Intervention

The need for hospitalization will be decided independently of the study by an on-duty physician in the emergency room. Whether hospitalized or not, the eligible children (rhinovirus positive wheezers, n=70) will be randomly assigned (2 separate randomization lists: one for hospitalized and one for out-patients) in a double-blind fashion to receive either oral prednisolone (first dose 2 mg/kg (max 60 mg), then 2 mg/kg/d (max 60 mg/d) in 3 divided doses for 3 days, Prednisolon®, 5 mg tablets, Oy Leiras Finland Ab, Helsinki, Finland) or placebo after informed consent had been obtained. The randomization code list will be stored in the hospital pharmacy and will be revealed only after all children had completed first 2 months of the study. Separate codes for each patients will be stored in patients charts and revealed in case of emergency. The tablets and packages will be indistinguishable in appearance from those of the active drug (Oy Leiras Finland Ab, Helsinki, Finland) and be provided in numbered containers. The study drugs will be administered by nurses independent of the study or by parents. The tablets will be minced and administered with jelly or yogurt. All patients will receive nebulized albuterol 0.15 mg/kg at 2 h intervals for the first 12 h, then at 4 h intervals while in the hospital. After discharge, beta2-agonists were used on demand. The patients will receive antibiotics or nebulized epinephrine (in emergency room or hospital) on demand.

Risk-benefit ratio

Previously, the efficacy of prednisolone has only been evaluated post-hoc in rhinovirus induced early wheezing in <3 year-old-children. The prevalence of relapses within 2 months after discharge was 22% in prednisolone group and 56% in placebo group. This observation needs to be confirmed in a prospective randomized trial, which is the purpose of the current study. Prednisolone has not been found beneficial in RSV-induced early wheezing in many studies and therefore, is not recommended to these children. Neither, prednisolone is used in upper respiratory tract infections without wheezing. Short courses (up to 5 days) of prednisolone have been used for decades in the treatment wheezing illnesses and they are well tolerated. There are no data that this dosage in this patient group could cause similar long-term neurological consequences as systemic corticosteroid treatment in mechanically ventilated premature infants suffering from severe respiratory distress syndrome.

Sample Size

Required sample size for the intervention will be >70 rhinovirus positive wheezing patients, which will include >35 infants for prednisolone group and >35 infants for placebo group. In addition, >200 healthy control children (no wheezing during the first 2 years of life) will be recruited and followed until school age.

Our primary endpoint is the occurrence of new wheezing episode within 2 months after discharge. According to our previous data on rhinovirus induced first or second episode of wheezing in children aged less than 3 years, the prevalence of relapses within 2 months after discharge in prednisolone group is 22% and in placebo group 56%. To maintain an alpha error of 0.05 and a beta error of 0.20, the required size of the sample is 29 children for each treatment group for the 2-month follow-up. When assessing the risk for the development of asthma at age 6 years, we expect 60% in the rhinovirus group and 18% in the RSV group to develop asthma by that age. We expect approximately 10-20% of the children to discontinue the study within 6 years. Thus, 35 children are needed in each group for the follow-up until school-age.

We expect approximately 15-25 subjects in each virus specific group to be sufficient to reveal immunologically or clinically meaningful differences.

Recruitment

Study subject will be recruited in the outpatient clinic of the Department of Pediatrics, or in the Pediatric Infectious Diseases Ward in the Turku University Hospital. Study physician/nurse or on-duty physician/nurse tells the guardian about the study and givens written information about the study. After the guardian has had adequate time the get familiar with the study and has had change to ask, his/her signature will be seeked to the informed consent form and the study will commence.

Description of Laboratory Methods for VINKU 2-study

The study protocol is presented in Table 1. Several laboratory analyses will enable us to address questions regarding the relationship between viral infections, T cell regulation, genetics, atopy, and pulmonary function. Laboratory work will be done according to modern standards.

Outcomes of the Intervention

Primary outcome: The occurrence of and time to a new physician-confirmed wheezing episode within 2 months after discharge; number of physician-confirmed wheezing episodes during the first 12 months after discharge; diagnoses of asthma during the full study period. Asthma is defined according to NAEPP Guidelines (http://www.nhlbi.nih.gov/guidelines/asthma).

Secondary outcomes: Up to 2 weeks after the acute respiratory tract infection, severity of symptoms (cough, wheeze, noisy breathing, breathlessness, rhinitis) will be assessed on a 4-graded scale (0-3, mild 1, moderate 2 and severe 3) by the parents as well as exact number of bronchodilator puffs used (symptom diary 1). Up to 2 months after the acute respiratory tract infection, parents will record days with rhinitis, cough, noisy breathing, wheezing, night-time symptoms, medication (bronchodilator, corticosteroid or antibiotics) and visits to physician or hospitalizations for wheezing (symptom diary 2). Up to 12 months, the number of out-patient care visits and hospitalizations for wheezing and courses of systemic or inhaled corticosteroids will be recorded (diary 3). Multiple immunologic markers and pulmonary function after 24-36 months and at age 6 years will be measured.

Termination of Study

Criteria for the termination of the study are:

1. Parent or guardian neglects the study orders.
2. Parent or guardian does not want to continue the study with any reason.
3. Completion of the study.

Ethical Aspects

The study protocol has been approved by the Ethics Committee of the Turku University Hospital in 11/2006 and will follow the rules of the current revision of the Declaration of Helsinki and the directives for clinical research by European Union (HE 20/2004). Patients or guardian won't get any financial benefits from the study. Children will be covered by the insurance (potilasvakuutus). This is an academic project and researchers have no conflicts of interests. Patient data will be confidential and won't be shared outside research group without coding. All deviations from the original protocol will be reported to the Ethics Committee of the Turku University Hospital and to the national authorities (Lääkelaitos).

Adverse events

All adverse events during hospitalization will be recorded on a four-point scale (0-3) and their possible relation to study drug will be assessed on a three-point scale (no, possible, likely, Appendix 4). Parents will be asked to record all adverse events on a two-week home symptom diary (Appendix 5). Investigator shall report all clinically meaningful adverse events in a timely correct manner to the national authorities (Lääkelaitos) according to national law, and to Leiras / Drug Safety Officer Johanna Kause. In case of premature termination of the trial, due to safety concerns, the investigator shall write a safety summary report and immediately forward this to Leiras and the national authorities. In case of an emergency, sealed envelope containing the randomization code will be available in the patient chart in the Turku University Hospital and can be easily opened.

ELIGIBILITY:
Inclusion Criteria:

* age 3-23 months
* be delivered at >=37 weeks
* first wheezing episode
* written informed consent from guardian

Exclusion Criteria:

* chronic illness other than atopy
* previous systemic or inhaled corticosteroid treatment
* participation to another study
* varicella contact if previously intact
* need for intensive care unit treatment, or
* poor understanding of Finnish

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2007-06; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of asthma | 1-7 years

SECONDARY OUTCOMES:
Home diary recordings for airway symptoms | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Pediatrics, Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Forsstrom V, Toivonen L, Homil K, Waris M, Pedersen CT, Bonnelykke K, Jartti T, Peltola V. Association of Asthma Risk Alleles With Acute Respiratory Tract Infections and Wheezing Illnesses in Young Children. J Infect Dis. 2023 Oct 18;228(8):990-998. doi: 10.1093/infdis/jiad075. PMID 36967681
- [Derived] Erkkola RA, Virta LJ, Vahlberg T, Jartti T. Prednisolone for the first rhinovirus induced wheezing reduces use of respiratory medication. Pediatr Allergy Immunol. 2022 Jan;33(1):e13668. doi: 10.1111/pai.13668. Epub 2021 Sep 29. No abstract available. PMID 34536305
- [Derived] Hurme P, Homil K, Lehtinen P, Turunen R, Vahlberg T, Vuorinen T, Camargo CA Jr, Gern JE, Jartti T. Efficacy of inhaled salbutamol with and without prednisolone for first acute rhinovirus-induced wheezing episode. Clin Exp Allergy. 2021 Sep;51(9):1121-1132. doi: 10.1111/cea.13960. Epub 2021 Jun 19. PMID 34062027
- [Derived] Koistinen A, Lukkarinen M, Turunen R, Vuorinen T, Vahlberg T, Camargo CA Jr, Gern J, Ruuskanen O, Jartti T. Prednisolone for the first rhinovirus-induced wheezing and 4-year asthma risk: A randomized trial. Pediatr Allergy Immunol. 2017 Sep;28(6):557-563. doi: 10.1111/pai.12749. Epub 2017 Aug 6. PMID 28660720
- [Derived] Lukkarinen M, Koistinen A, Turunen R, Lehtinen P, Vuorinen T, Jartti T. Rhinovirus-induced first wheezing episode predicts atopic but not nonatopic asthma at school age. J Allergy Clin Immunol. 2017 Oct;140(4):988-995. doi: 10.1016/j.jaci.2016.12.991. Epub 2017 Mar 25. PMID 28347734
- See also: home page of the VINKU study group — http://vinku.utu.fi/